CLINICAL TRIAL: NCT04046770
Title: Innovative Device for Intravenous Administration
Acronym: SeringaDUO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Escola Superior de Enfermagem de Coimbra (Other)
Collaborators: Hospital de Braga (Other); Unidade Local de Saúde de Coimbra, EPE (Other); Hospital Distrital da Figueira da Foz, EPE (Unknown)
Responsible Party: Principal Investigator, Pedro Miguel Santos Dinis Parreira, Ph.D, Coordinating Professor, Escola Superior de Enfermagem de Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SeringaDuo
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Safety Issues; Medical Device
Keywords: safety; Effectiveness; Double-chamber syringe; Clinical research; medical devices; nurses; hospital setting

STUDY DESIGN:
Intervention Model Description: A multi-centre, two-arm randomised controlled trial with partially blinded outcome assessment, of 146 adult patients. After eligibility analysis and informed consent, participants will receive usual intravenous administration of drugs with subsequent flushing procedures, with the double-chamber syringe (arm A) or with the classical syringes (arm B). The outcomes assessment will be performed on a daily basis by the unblind research team, with the same procedures in both groups. Some main outcomes, such as phlebitis and infiltration, will also be evaluated by nurses from a blind research team and registered once a day.
Masking Description: Patients and clinical staff will not be entirely blind after group allocation due to the nature of the interventions. Despite this, participants will not be directly informed of their group allocation in terms of usual care or intervention, and the nurses in the clinical staff will only be informed about the broad purposes of the research [41] - the study of a new double-chamber syringe for intravenous administration and flushing. In contrast, research nurses from the team outside the orthopaedic department will be blinded when rating some of the main outcomes such as phlebitis and infiltration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-Chamber Syringe (Experimental): Intravenous administration of drugs and flushing with the Double-Chamber Syringe
  Interventions: Device: Drug administration and Flushing procedure using Double-Chamber Syringe
- Classical Syringes (Active Comparator): Intravenous administration of drugs and flushing with the classical syringe
  Interventions: Device: Drug administration and Flushing procedure using Classic Syringe

INTERVENTIONS:
Device: Drug administration and Flushing procedure using Double-Chamber Syringe — The new device will allow the professional to conduct all the procedure (assure the patency/enables the pre-flushing), drugs administration and flushing, using only one device.
  Arms: Double-Chamber Syringe
Device: Drug administration and Flushing procedure using Classic Syringe — To fully complete the intravenous drug administration with rigor, nurses should flush the catheter pre, post and inbetween drug administration. This implies the use of two or three syringes.
  Arms: Classical Syringes

SUMMARY:
The prevention of catheter-related complications is nowadays an important topic of research. Flushing the catheters is considered an important clinical procedure in preventing malfunction and several complications such as phlebitis or infection. Considering the latest guidelines of the Infusion Nurses Society, the flushing involves a pre and post-drug administration, requiring different syringes (with associated overall increased times of preparation/administration of intravenous medication by nurses, also increasing the need for manipulation of the venous catheter).

A multi-centre, two-arm randomised controlled trial with partially blinded outcome assessment, of 146 adult patients. After eligibility analysis and informed consent, participants will receive usual intravenous administration of drugs with subsequent flushing procedures, with the double-chamber syringe (arm A) or with the classical syringes (arm B). The outcomes assessment will be performed on a daily basis by the unblind research team, with the same procedures in both groups. Some main outcomes, such as phlebitis and infiltration, will also be evaluated by nurses from a blind research team and registered once a day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years or above, admitted to the orthopaedic department;
* Patients with the ability to fully communicate in Portuguese;
* Patients able to consent;
* Prescribed PIVC for intravenous therapeutic administration;
* PIVC expected to remain for at least 24 hours;
* PIVC inserted at the orthopaedic department;
* PIVC size 18 gauge (G) or 20 G;
* Anatomical insertion site in arm, forearm, or back of the hand;
* PIVC secured with a transparent, semi-permeable polyurethane film dressing.

Exclusion Criteria:

* - Patients with a known infectious disease;
* Patients with leucocytosis, defined as ≥1200 leukocytes/mm3;
* Patients with anaemia, with haemoglobin levels <13g/dl for men, and <12g/dl for women;
* Patients receiving immunosuppressive treatment within 6 months prior to hospital admission;
* Patients receiving chemotherapy or radiotherapy within 6 months prior to hospital admission;
* Patients with body mass index below 16 kg/m2 or above 39 kg/m2;
* Anatomical insertion site in flexion areas (e.g. cubital fossa region) or lower members;
* Skin lesions at the insertion site (e.g. previous infiltration, dermatitis, burns) and skin alterations such as tattoos;
* Peripheral venous alterations resulting from previous hospital admissions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Catheter-related complications: phlebitis | This outcome will be assessed during the patient's hospital stay (through study completion, an average of 9 months) and 48 hours to 72 hours after catheter removal.
  Phlebitis (the irritation or inflammation to the vein wall, associated with warmth, tenderness, erythema or palpable cord) is the most frequent PIVC-related complication, which may have mechanical, chemical, or bacterial causes
Catheter-related complications: infiltration | This outcome will be assessed during the patient's hospital stay (through study completion, an average of 9 months).
  Moreover, the extravasation or infiltration of fluids may be responsible for local oedema due to the pervasion of intravenous fluid into the interstitial compartment, causing inflammation of the tissue around the catheter site.
Catheter-related complications: occlusion | This outcome will be assessed during the patient's hospital stay (through study completion, an average of 9 months).
  Occlusion is defined as any circumstance in which the Peripheral Intravenous Catheter (PIVC) does not enable to flush the catheter or infuse fluids/medications and it is a clinical sign of catheter malfunctioning

SECONDARY OUTCOMES:
Other catheter-related removal causes not related with the primary outcomes | This outcome will be assessed during the patient's hospital stay (through study completion, an average of 9 months) and in 48 hours to 72 hours after catheter removal.
  The secondary outcomes involve other reasons for catheter removal (e.g. accidental dislodgment), maintenance time of the catheter, number of syringes and catheters used during the intravenous treatment, catheterization attempts, nurses' perception about risk and safety, as well as the satisfaction of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Parreira, PhD, Principal Investigator — Coordinating Professor

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.

REFERENCES:
- [Background] Chopra V, Flanders SA, Saint S, Woller SC, O'Grady NP, Safdar N, Trerotola SO, Saran R, Moureau N, Wiseman S, Pittiruti M, Akl EA, Lee AY, Courey A, Swaminathan L, LeDonne J, Becker C, Krein SL, Bernstein SJ; Michigan Appropriateness Guide for Intravenouse Catheters (MAGIC) Panel. The Michigan Appropriateness Guide for Intravenous Catheters (MAGIC): Results From a Multispecialty Panel Using the RAND/UCLA Appropriateness Method. Ann Intern Med. 2015 Sep 15;163(6 Suppl):S1-40. doi: 10.7326/M15-0744. PMID 26369828
- [Background] Abolfotouh MA, Salam M, Bani-Mustafa A, White D, Balkhy HH. Prospective study of incidence and predictors of peripheral intravenous catheter-induced complications. Ther Clin Risk Manag. 2014 Dec 8;10:993-1001. doi: 10.2147/TCRM.S74685. eCollection 2014. PMID 25525365
- [Background] Braga LM, Parreira PM, Oliveira ASS, Monico LDSM, Arreguy-Sena C, Henriques MA. Phlebitis and infiltration: vascular trauma associated with the peripheral venous catheter. Rev Lat Am Enfermagem. 2018;26:e3002. doi: 10.1590/1518-8345.2377.3002. Epub 2018 May 17. PMID 29791668
- [Background] Ho KH, Cheung DS. Guidelines on timing in replacing peripheral intravenous catheters. J Clin Nurs. 2012 Jun;21(11-12):1499-506. doi: 10.1111/j.1365-2702.2011.03974.x. Epub 2012 Feb 17. PMID 22340078
- [Background] Park SM, Jeong IS, Kim KL, Park KJ, Jung MJ, Jun SS. The Effect of Intravenous Infiltration Management Program for Hospitalized Children. J Pediatr Nurs. 2016 Mar-Apr;31(2):172-8. doi: 10.1016/j.pedn.2015.10.013. Epub 2015 Nov 19. PMID 26608556
- [Background] Rickard CM, McCann D, Munnings J, McGrail MR. Routine resite of peripheral intravenous devices every 3 days did not reduce complications compared with clinically indicated resite: a randomised controlled trial. BMC Med. 2010 Sep 10;8:53. doi: 10.1186/1741-7015-8-53. PMID 20831782
- [Background] Martinez JA, Piazuelo M, Almela M, Blecua P, Gallardo R, Rodriguez S, Escalante Z, Robau M, Trilla A. Evaluation of add-on devices for the prevention of phlebitis and other complications associated with the use of peripheral catheters in hospitalised adults: a randomised controlled study. J Hosp Infect. 2009 Oct;73(2):135-42. doi: 10.1016/j.jhin.2009.06.031. Epub 2009 Aug 27. PMID 19712998
- [Background] Wallis MC, McGrail M, Webster J, Marsh N, Gowardman J, Playford EG, Rickard CM. Risk factors for peripheral intravenous catheter failure: a multivariate analysis of data from a randomized controlled trial. Infect Control Hosp Epidemiol. 2014 Jan;35(1):63-8. doi: 10.1086/674398. Epub 2013 Dec 2. PMID 24334800
- [Background] Capdevila JA, Guembe M, Barberan J, de Alarcon A, Bouza E, Farinas MC, Galvez J, Goenaga MA, Gutierrez F, Kestler M, Llinares P, Miro JM, Montejo M, Munoz P, Rodriguez-Creixems M, Sousa D, Cuenca J, Mestres CA; on behalf the SEICAV, SEMI, SEQ and SECTCV Societies. 2016 Expert consensus document on prevention, diagnosis and treatment of short-term peripheral venous catheter-related infections in adult. Rev Esp Quimioter. 2016 Aug;29(4):230-8. Epub 2016 Aug 28. PMID 27580009
- [Background] Loveday HP, Wilson JA, Pratt RJ, Golsorkhi M, Tingle A, Bak A, Browne J, Prieto J, Wilcox M, UK Department of Health. epic3: national evidence-based guidelines for preventing healthcare-associated infections in NHS hospitals in England. J Hosp Infect. 2014 Jan;86 Suppl 1:S1-70. doi: 10.1016/S0195-6701(13)60012-2. PMID 24330862
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee (HICPAC). Guidelines for the prevention of intravascular catheter-related infections. Clin Infect Dis. 2011 May;52(9):e162-93. doi: 10.1093/cid/cir257. Epub 2011 Apr 1. No abstract available. PMID 21460264
- [Background] Marsh N, Webster J, Mihala G, Rickard CM. Devices and dressings to secure peripheral venous catheters to prevent complications. Cochrane Database Syst Rev. 2015 Jun 12;2015(6):CD011070. doi: 10.1002/14651858.CD011070.pub2. PMID 26068958
- [Background] Goossens GA. Flushing and Locking of Venous Catheters: Available Evidence and Evidence Deficit. Nurs Res Pract. 2015;2015:985686. doi: 10.1155/2015/985686. Epub 2015 May 14. PMID 26075094
- [Background] Keogh S, Flynn J, Marsh N, Higgins N, Davies K, Rickard CM. Nursing and midwifery practice for maintenance of vascular access device patency. A cross-sectional survey. Int J Nurs Stud. 2015 Nov;52(11):1678-85. doi: 10.1016/j.ijnurstu.2015.07.001. Epub 2015 Jul 11. PMID 26206327
- [Background] Ferroni A, Gaudin F, Guiffant G, Flaud P, Durussel JJ, Descamps P, Berche P, Nassif X, Merckx J. Pulsative flushing as a strategy to prevent bacterial colonization of vascular access devices. Med Devices (Auckl). 2014 Nov 7;7:379-83. doi: 10.2147/MDER.S71217. eCollection 2014. PMID 25404862
- [Background] Bishop L, Dougherty L, Bodenham A, Mansi J, Crowe P, Kibbler C, Shannon M, Treleaven J. Guidelines on the insertion and management of central venous access devices in adults. Int J Lab Hematol. 2007 Aug;29(4):261-78. doi: 10.1111/j.1751-553X.2007.00931.x. PMID 17617077
- [Background] Guiffant G, Durussel JJ, Merckx J, Flaud P, Vigier JP, Mousset P. Flushing of intravascular access devices (IVADs) - efficacy of pulsed and continuous infusions. J Vasc Access. 2012 Jan-Mar;13(1):75-8. doi: 10.5301/JVA.2011.8487. PMID 21748725
- [Background] Ngo A, Murphy S. A theory-based intervention to improve nurses' knowledge, self-efficacy, and skills to reduce PICC occlusion. J Infus Nurs. 2005 May-Jun;28(3):173-81. doi: 10.1097/00129804-200505000-00005. PMID 15912072
- [Background] Boutron I, Guittet L, Estellat C, Moher D, Hrobjartsson A, Ravaud P. Reporting methods of blinding in randomized trials assessing nonpharmacological treatments. PLoS Med. 2007 Feb;4(2):e61. doi: 10.1371/journal.pmed.0040061. PMID 17311468
- [Background] Keogh S, Flynn J, Marsh N, Mihala G, Davies K, Rickard C. Varied flushing frequency and volume to prevent peripheral intravenous catheter failure: a pilot, factorial randomised controlled trial in adult medical-surgical hospital patients. Trials. 2016 Jul 26;17(1):348. doi: 10.1186/s13063-016-1470-6. PMID 27456005
- [Background] Marsh N, Webster J, Flynn J, Mihala G, Hewer B, Fraser J, Rickard CM. Securement methods for peripheral venous catheters to prevent failure: a randomised controlled pilot trial. J Vasc Access. 2015 May-Jun;16(3):237-44. doi: 10.5301/jva.5000348. Epub 2015 Feb 4. PMID 25656258
- [Background] Rickard CM, Webster J, Wallis MC, Marsh N, McGrail MR, French V, Foster L, Gallagher P, Gowardman JR, Zhang L, McClymont A, Whitby M. Routine versus clinically indicated replacement of peripheral intravenous catheters: a randomised controlled equivalence trial. Lancet. 2012 Sep 22;380(9847):1066-74. doi: 10.1016/S0140-6736(12)61082-4. PMID 22998716
- [Background] Tuffaha HW, Rickard CM, Webster J, Marsh N, Gordon L, Wallis M, Scuffham PA. Cost-effectiveness analysis of clinically indicated versus routine replacement of peripheral intravenous catheters. Appl Health Econ Health Policy. 2014 Feb;12(1):51-8. doi: 10.1007/s40258-013-0077-2. PMID 24408785
- [Background] Dillon MF, Curran J, Martos R, Walsh C, Walsh J, Al-Azawi D, Lee CS, O'Shea D. Factors that affect longevity of intravenous cannulas: a prospective study. QJM. 2008 Sep;101(9):731-5. doi: 10.1093/qjmed/hcn078. Epub 2008 Jul 11. PMID 18621805
- [Background] Dunda SE, Demir E, Mefful OJ, Grieb G, Bozkurt A, Pallua N. Management, clinical outcomes, and complications of acute cannula-related peripheral vein phlebitis of the upper extremity: A retrospective study. Phlebology. 2015 Jul;30(6):381-8. doi: 10.1177/0268355514537254. Epub 2014 May 20. PMID 24844248
- [Derived] Parreira P, Sousa LB, Marques IA, Santos-Costa P, Braga LM, Cruz A, Salgueiro-Oliveira A. Double-chamber syringe versus classic syringes for peripheral intravenous drug administration and catheter flushing: a study protocol for a randomised controlled trial. Trials. 2020 Jan 14;21(1):78. doi: 10.1186/s13063-019-3887-1. PMID 31937342